CLINICAL TRIAL: NCT00003067
Title: Intracavitary Interleukin-2 (IL-2) and Lymphokine-Activated Killer (LAK) Cell Therapy for Malignant Gliomas
Brief Title: Biological Therapy in Treating Patients With Primary or Advanced Glioma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065739; NYWCCC-0902499; NYWCCC-IMMUNE-0902499; SIUH-RP-96-004; NCI-V97-1326
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2008-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Glioma; Gliosarcoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: lymphokine-activated killer cells

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells in patients with primary or advanced glioma.

PURPOSE: Clinical trial to study the effectiveness of biological therapy with interleukin-2 and lymphokine-activated killer cells in treating patients who have primary, recurrent, or refractory malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Confirm the antitumor efficacy of intracavitary interleukin-2 plus autologous lymphokine-activated killer cells in patients with primary, recurrent or refractory malignant gliomas.
* Determine whether the induction of a regional, intracavitary, eosinophilia is a prognosticator of response to immunotherapy and long term survival in these patients.

OUTLINE: Patients receive cytoreductive tumor surgery and/or biopsy and implantation of intracavitary Ommaya reservoir prior to therapy induction.

Patients undergo outpatient leukapheresis on day -4 or -5, and cells are incubated ex vivo with interleukin-2 (IL-2). Lymphokine-activated killer (LAK) cells and IL-2 are infused on day 1. Bolus infusions of low-dose IL-2 are administered on days 3, 5, 8, 10, and 12, followed by a rest period on days 13-24. The course is repeated on day 25 starting with leukapheresis. Therapy courses are repeated for up to 1 year for stable disease or response to therapy. Maintenance doses repeat every 4-6 months thereafter.

Disease restaging is done every 8-12 weeks.

PROJECTED ACCRUAL: A total of 30 patients per year will be enrolled.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or radiographically proven primary, recurrent, or refractory malignant gliomas (glioblastoma, anaplastic astrocytoma, and mixed anaplastic glioma)

  * Must be a candidate for neurosurgical biopsy or tumor debulking

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance Status:

* Karnofsky 60-100%

Life Expectancy:

* Greater than 4 months

Hematopoietic:

* Granulocytes greater than 1,500/mm^3
* Platelet count greater than 50,000/mm^3
* PT and PTT within normal limits

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal

Renal:

* Creatinine less than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No congestive heart failure
* No coronary artery disease
* No serious cardiac arrhythmias
* No prior myocardial infarction

Pulmonary:

* No major pulmonary problems

Other:

* No history of neurologic disease (except related to brain tumor)
* No psychosis
* No impaired cognitive function
* No significant concurrent medical illness
* No active infection requiring antibiotic therapy
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate peripheral veins to permit leukapheresis, or placement of indwelling central vascular access device
* No hepatitis B or C
* HIV negative
* No prior autoimmune disease
* Allergy to gentamicin is allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 weeks since prior immunotherapy and recovered
* No concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for carmustine) and recovered
* No concurrent chemotherapy

Endocrine therapy:

* Reduction or elimination of corticosteroids
* Not greater than 0.15 mg/kg/day dexamethasone equivalent

Radiotherapy:

* At least 6 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* Prior surgery is allowed

Other:

* Concurrent therapy with acetaminophen, anticonvulsant agents, and headache pain medications is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-07

CONTACTS AND LOCATIONS:
Overall Officials: Roberta L. Hayes, PhD, Study Chair — Immune Therapy, LLC
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

REFERENCES:
- [Result] Hayes RL, Koslow M, Hiesiger EM, Hymes KB, Hochster HS, Moore EJ, Pierz DM, Chen DK, Budzilovich GN, Ransohoff J. Improved long term survival after intracavitary interleukin-2 and lymphokine-activated killer cells for adults with recurrent malignant glioma. Cancer. 1995 Sep 1;76(5):840-52. doi: 10.1002/1097-0142(19950901)76:53.0.co;2-r. PMID 8625188